CLINICAL TRIAL: NCT01034462
Title: A Double-blind, Placebo-Controlled, Flexible-Dose Study of F2695 SR in Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of Levomilnacipran ER (F2695 SR) in Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LVM-MD-03
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Levomilnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Levomilnacipran ER capsules, flexible dose, oral administration, once daily dosing.
  Interventions: Drug: Levomilnacipran ER
- 2 (Placebo Comparator): Matching placebo capsules, oral administration, once daily dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levomilnacipran ER — Levomilnacipran ER capsules, flexible dose, oral administration, once daily dosing. Study drug is to be given orally, in capsule form, once daily, for 8 weeks
  Arms: 1
Drug: Placebo — Matching placebo to be given orally, in capsule form, once daily, for 8 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of Levomilnacipran ER versus placebo in the treatment of outpatients with major depressive disorder

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-80 years old
* Currently meet the DSM-IV-TR criteria for Major Depressive Disorder
* The patient's current depressive episode must be at least 4 weeks in duration

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women with childbearing potential who are not practicing a reliable method of birth control.
* Patients with a history of meeting DSM-IV-TR criteria for: a. any manic or hypomanic episode; b. schizophrenia or any other psychotic disorder; c. obsessive-compulsive disorder.
* Patients who are considered a suicide risk

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Gommoll, MS, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories Inc.
Locations (23):
- United States (23):
  - Forest Investigative Site 055, Dothan, Alabama
  - Forest Investigative Site 065, Highlands Ranch, Colorado
  - Forest Investigative Site 057, Boca Raton, Florida
  - Forest Investigative Site 060, Boca Raton, Florida
  - Forest Investigative Site 064, Gainesville, Florida
  - Forest Investigative Site 053, Ocala, Florida
  - Forest Investigative Site 061, Orlando, Florida
  - Forest Investigative Site 059, Winter Park, Florida
  - Forest Investigative Site 070, Atlanta, Georgia
  - Forest Investigative Site 066, Smyrna, Georgia
  - Forest Investigative Site 072, Chicago, Illinois
  - Forest Investigative Site 050, Oak Brook, Illinois
  - Forest Investigative Site 063, Indianapolis, Indiana
  - Forest Investigative Site 071, Prairie Village, Kansas
  - Forest Investigative Site 052, Shreveport, Louisiana
  - Forest Investigative Site 051, Brooklyn, New York
  - Forest Investigative Site 056, Oklahoma City, Oklahoma
  - Forest Investigative Site 067, Oklahoma City, Oklahoma
  - Forest Investigative Site 058, Salem, Oregon
  - Forest Investigative Site 054, Allentown, Pennsylvania
  - Forest Investigative Site 062, San Antonio, Texas
  - Forest Investigative Site 068, Virginia Beach, Virginia
  - Forest Investigative Site 069, Spokane, Washington

REFERENCES:
- [Derived] Wesnes KA, Gommoll C, Chen C, Sambunaris A, McIntyre RS, Harvey PD. Effects of levomilnacipran extended-release on major depressive disorder patients with cognitive impairments: post-hoc analysis of a phase III study. Int Clin Psychopharmacol. 2017 Mar;32(2):72-79. doi: 10.1097/YIC.0000000000000157. PMID 27861191
- [Derived] Cutler AJ, Gommoll CP, Chen C, Greenberg WM, Ruth A. Levomilnacipran Extended-Release Treatment in Patients With Major Depressive Disorder: Improvements in Functional Impairment Categories. Prim Care Companion CNS Disord. 2015 Jun 11;17(3):10.4088/PCC.14m01753. doi: 10.4088/PCC.14m01753. eCollection 2015. PMID 26644957
- [Derived] Sambunaris A, Bose A, Gommoll CP, Chen C, Greenberg WM, Sheehan DV. A phase III, double-blind, placebo-controlled, flexible-dose study of levomilnacipran extended-release in patients with major depressive disorder. J Clin Psychopharmacol. 2014 Feb;34(1):47-56. doi: 10.1097/JCP.0000000000000060. PMID 24172209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited over a 21-month period from December of 2009 to September of 2011 at 23 studies sites in the United States.
Pre-assignment Details: Patients went through a 1-week single-blind placebo run-in period immediately preceding an 8-week double-blind treatment period.
Groups:
- Placebo: Matching placebo capsules, oral administration, once daily dosing for 8 weeks.
- Levomilnacipran ER: Levomilnacipran ER capsules, flexible dose, oral administration, once daily dosing for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Levomilnacipran ER
Started | 217 | 217
Completed | 172 | 163
Not Completed | 45 | 54
Not completed — Adverse Event | 7 | 17
Not completed — Lack of Efficacy | 4 | 4
Not completed — Protocol Violation | 10 | 7
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Lost to Follow-up | 14 | 16
Not completed — Other reasons | 1 | 2

BASELINE CHARACTERISTICS:
Population: While 442 patients were randomized to receive double-blind treatment, 8 of these patients discontined before receiving double-blind treatment. The Baseline Participant population is based on the 434 randomized patients who went on to receive double-blind treatment (Safety Population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Levomilnacipran ER | Total
Number analyzed (Participants) | 217 | 217 | 434
Age Continuous [Mean (Standard Deviation); unit: years] | 44.6 (13.9) | 45.0 (13.2) | 44.8 (13.5)
Age, Customized [Number; unit: participants]
  18 years to 19 years | 2 | 2 | 4
  20 years to 29 years | 38 | 34 | 72
  30 years to 39 years | 37 | 44 | 81
  40 years to 49 years | 51 | 40 | 91
  50 years to 59 years | 57 | 68 | 125
  60 years to 80 years | 32 | 29 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 140 | 283
  Male | 74 | 77 | 151
Race/Ethnicity, Customized [Number; unit: participants]
  White | 182 | 177 | 359
  Black or African American | 28 | 33 | 61
  Asian | 2 | 2 | 4
  American Indian or Alaska native | 1 | 1 | 2
  Other | 4 | 4 | 8
  Hispanic or Latino | 17 | 21 | 38
  Not Hispanic or Latino | 200 | 196 | 396
Region of Enrollment [Number; unit: participants]
  United States | 217 | 217 | 434
Weight [Mean (Standard Deviation); unit: kg] | 84.58 (18.15) | 84.47 (18.98) | 84.52 (18.55)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms Per Meter Squared] | 29.60 (5.30) | 29.20 (5.45) | 29.40 (5.37)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: MADRS was used to assess depressive symptomatology during the past week. Patients are rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest.
  Each item of the 10 items are scored on a 7-point scale. A score of 0 indicates the absence of symptoms,and a score of 6 indicates symptoms of maximum severity. The total MADRS score for this measure ranges from 0 (absence of symptoms) to 60 (maximum severity).
Time Frame: From Baseline to Week 8
Population: The Safety Population consisted of 434 randomized patients who took at least 1 dose of double-blind investigational product. The Intent-to-Treat (ITT) Population consisted 429 patients in the Safety Population who had at least 1 postbaseline assessment of the MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Matching placebo capsules, oral administration, once daily dosing.
  Placebo : Matching placebo to be given orally, in capsule form, once daily, for 8 weeks.
Arm/Group | Placebo | Levomilnacipran ER
Number analyzed (Participants) | 214 | 215
units on a scale | -12.2 (0.78) | -15.3 (0.79)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -3.095, 95% CI 2-sided [-5.256 to -0.935]

2. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale (SDS) is a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point continuum (0 = no impairment to 10 = most severe) with the total SDS score ranging from 0 (no impairment) to 30 (most severe)
Time Frame: From Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Levomilnacipran ER
Number analyzed (Participants) | 214 | 215
units on a scale | -5.4 (0.57) | -8.0 (0.58)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran ER; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -2.632, 95% CI 2-sided [-4.193 to -1.070]

ADVERSE EVENTS:
Time Frame: Adverse event data was collection over a 25-month period from December 2009 to January 2012 at 23 study sites in the U.S.
Description: The Serious Adverse Event data presented here is for the safety population. The Other Adverse Event data presented here is for the safety population during the 8 week double-blind treatment period.
Arm/Group | Placebo | Levomilnacipran ER
Serious Adverse Events (participants affected / at risk) | 3/217 | 4/217
Other Adverse Events (participants affected / at risk) | 79/217 | 151/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=217) | Levomilnacipran ER (N=217)
Non-cardiac chest pain (General disorders) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=217) | Levomilnacipran ER (N=217)
Nausea (Nervous system disorders) | 8 | 47
Headache (Nervous system disorders) | 27 | 38
Dizziness (Nervous system disorders) | 7 | 28
Dry mouth (Gastrointestinal disorders) | 24 | 27
Constipation (Gastrointestinal disorders) | 8 | 22
Tachycardia (Cardiac disorders) | 6 | 18
Urinary hesitation (Renal and urinary disorders) | 0 | 17
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 15
Insomnia (Psychiatric disorders) | 5 | 15
Diarrhoea (Gastrointestinal disorders) | 12 | 14
Vomiting (Gastrointestinal disorders) | 2 | 14
Upper respiratory tract infection (Infections and infestations) | 9 | 13
Hypertension (Vascular disorders) | 3 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.